CLINICAL TRIAL: NCT02158780
Title: Expertise-Based Randomized Controlled Trial of Scrotal Versus Inguinal (Standard) Orchidopexy on Postoperative Pain: EXPRESSO Trial
Brief Title: Expertise-Based Randomized Controlled Trial of Scrotal Versus Inguinal Orchidopexy on Post-operative Pain
Acronym: EXPRESSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: McMaster Surgical Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EXPRESSO
Record Dates: First submitted 2014-05-20; First posted 2014-06-09 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2019-08

CONDITIONS: Low-lying Unilateral Palpable Undescended Testis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Scrotal Orchidopexy (Experimental): Single incision
  Interventions: Procedure: Scrotal Orchidopexy
- Inguinal Orchidopexy (Other): Double Incision (Standard)
  Interventions: Procedure: Inguinal Orchidopexy

INTERVENTIONS:
Procedure: Scrotal Orchidopexy — Single incision
  Arms: Scrotal Orchidopexy
Procedure: Inguinal Orchidopexy — Double Incision (Standard)
  Arms: Inguinal Orchidopexy

SUMMARY:
Undescended Testis is the most common congenital abnormality of the genitalia in boys and it is commonly managed by surgical intervention. Evidence in the medical literature to support the superiority of either scrotal or inguinal (standard) orchidopexy is lacking. To determine which technique is superior, this study focuses on the degree of post-operative pain after surgery. Therefore, the objective of this randomized control trial is to determine if scrotal orchidopexy reduces postoperative pain in children diagnosed with undescended testis when compared to standard inguinal orchidopexy.

DETAILED DESCRIPTION:
Undescended Testis is the most common congenital abnormality of the genitalia in boys and it is commonly managed by surgical intervention. Evidence in the medical literature to support the superiority of either scrotal or inguinal (standard) orchidopexy is lacking. To determine which technique is superior, this study focuses on the degree of post-operative pain after surgery. Therefore, the objective of this randomized control trial is to determine if scrotal orchidopexy reduces postoperative pain in children diagnosed with undescended testis when compared to standard inguinal orchidopexy. At the first pre-operative clinic visit participating paediatric urologist will diagnose patients with low-lying palpable UDT. Patients who meet eligibility criteria will be invited to participate in this trial. A computer generated randomization list will be created using random blocks of multiple sizes (4, 6 and 8), by the McMaster Paediatric Surgery Research Collaborative's web-based randomization system. Patients will be allocated to intervention (scrotal orchidopexy) or control (standard inguinal orchidopexy) groups by logging in to the secure central randomization website. Patients will be stratified and randomized by centre into a 1:1 parallel allocation ratio.Primary Outcome: Post-operative pain during recovery phase Sample size calculated using single primary outcome of analgesic use. However, pain will also be measured in alternative ways using pain scales as a secondary outcome. Analgesic use post-operatively (during hospital stay): Defined as the number of doses and total consumption of morphine (standardized dose of 0.2 mg/kg/dose orally or 0.02 to 0.1 mg/kg/dose IV) or oral acetaminophen (15mg/kg/dose) or Ibuprofen (10mg/kg/dose) administered by PACU and SDSU nurses following surgery. Analgesic use post-discharge: Defined as number of standardized doses and total consumption of acetaminophen (15 mg/kg/dose) and Ibuprofen (10 mg/kg/dose) administered by parent/guardian at home post-discharge.Secondary Outcomes: Duration of surgery, Pain Scores, Success rate, Complications. Duration of surgery (min): Defined as time beginning when anesthesia is ready until patient is moved to PACU. Recorded on patient discharge sheet by study nurse. Time to discharge: Defined as duration of time from entering PACU to readiness to discharge from PACU or same day-surgery unit (if applicable). Recording by study nurse on discharge sheet. Pain Scales post-operative:Mean of highest pain score in each patient: Self-reported pain scales are gold-standard for reporting pain; however, since this study sample comprises of pre-verbal children, an observer pain tool will be used. Specifically, pain scores will be measured through a reliable and validated observer-rated Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) and Face, Legs, Activity, Cry, Consolability (FLACC) Behavioural Scale30 by two trained, blinded, and independent study personnel. Both study personnel will measure pain at admission and discharge during the recovery phase. Recovery phase is defined as post-operative period in the post-anesthesia care unit (PACU) and same day surgery unit (SDSU). Patients usually recover for an average of two hours before being discharged. Highest pain score will be determined by blinded analysts. At monthly intervals, inter-rater reliability between study personnel will be assessed and re-trained to ensure high consistency in score ratings.

Mean overall pain sore: Average pain score (standard deviation) throughout recovery phase. Pain scales post-discharge: Information measured at home by parent/guardian. Collected by study personnel at 24 hour follow-up telephone call. Mean of the highest pain score in each patient: Assessed through validated and reliable Parents Postoperative Pain Measure (PPPM)and Toddler-Preschooler Postoperative Pain Scale (TPPPS) by trained and parent/guardian 24 hrs post-discharge. Complication rate: Defined as number of complications per group. Complications include surgical site infection, scrotal hematoma, bleeding, scrotal swelling, hernia formation, testicular atrophy, and wound dehiscence. Assessed 6-8 weeks post-surgery by a trained clinician who was not involved in administering surgery for this study. Success rate of procedure: Defined as number of testis successfully lowered into the lower scrotum at a 6-8 week follow-up visit evaluated by a trained clinician.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis with palpable undescended testis (or testes);
2. Child is between 10 mos - 7 years of age;
3. Child requires either scrotal or inguinal orchidopexy

Exclusion Criteria

1. Laparoscopic surgery for intra-abdominal testis or peeping testis (carnalicular);
2. Child underwent previous orchidopexy surgery

Ages: 10 Months to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 162 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
Analgesic use post-operatively (during hospital stay) | Measured dosage post-surgery (on average 45 minutes later)
  Defined as the number of doses of morphine (standardized dose of 0.2 mg/kg) or Tylenol (15mg/kg) or Ibuprofen (10mg/kg) administered by PACU and SDSU nurses following surgery.
Analgesic use post-discharge | Measure at 6 hour intervals post discharge for 48 hours
  Defined as number of standardized doses of Tylenol (15 mg/kg) and Ibuprofen (10 mg/kg) administered by parent/guardian at home post-discharge.

SECONDARY OUTCOMES:
Pain Scales post-operative (during hospital stay) | Measure at patient admission and discharge at 30 minute intervals.
  Pain scores will be measured through a reliable and validated observer-rated Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) by two trained, blinded, and independent study personnel. Both study personnel will measure pain at admission and discharge during the recovery phase.
Pain Scales post-operative (during hospital stay) | Measure at patient admission and discharge at 30 minute intervals.
  Pain scores will be measured through a reliable and validated observer-rated Face, Legs, Activity, Cry, Consolability (FLACC) Behavioural Scale by two trained, blinded, and independent study personnel. Both study personnel will measure pain at admission and discharge during the recovery phase.
Pain scales post-discharge | Measure at 6 hour intervals post discharge for 48 hours
  Assessed through validated and reliable Parents Postoperative Pain Measure (PPPM) by trained and blinded parent/guardian at 6, 12,18, 24, 30, 36, 42, 48 hrs post-discharge
Analgesic use | Measured dosage at the beginning of surgery and post-surgery (on average 45minutes later)
  Amount of pain medication administered to patient intra and post operatively
Duration of surgery (min) | Record duration of operative time (takes on average 30-45 minutes)
  Obtained from operative case notes. Defined as beginning of first skin incision and ending when post-operative dressing has been applied.
Time to discharge | Duration of time from being admitted for surgery until time discharged (which is on average 4 hours)
  Defined as duration of time from entering PACU to discharge from day-surgery unit. Recording by study nurse on discharge sheet.
Short term complications | Measured at 48 hour follow-up clinic visit
  Examples include surgical site infection, scrotal hematoma, bleeding, scrotal swelling and wound dehiscence
Long-term complications | Measured at 3 and 6 month follow-up clinic visit
  Examples include: hernia formation and testicular atrophy
Success rate | Measured at 3 month followup clinic visit
  Success rate in this study is defined by the number of viable testicles successfully positioned into the lower part of the scrotum.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Braga, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster Children Hospital, Hamilton, Ontario, Canada